CLINICAL TRIAL: NCT03578887
Title: A Twin Study of Obesity Pathogenesis Using fMRI
Brief Title: A Cohort Study of Weight Loss and Gliosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Ellen Schur, MD, MS, Assistant Professor, School of Medicine: General Internal Medicine, University of Washington
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00002978; 2R01DK089036-06 (NIH); 1K24HL144917-01A1 (NIH)
Record Dates: First submitted 2018-06-25; First posted 2018-07-06 (Actual); Results first posted 2025-07-28 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Obesity, Gliosis, Weight-Loss
Keywords: Obesity, Gliosis, Weight-Loss, Roux-en-Y Gastric Bypass, Type 2 Diabetes Mellitus
MeSH Terms: conditions — Obesity; Gliosis; Weight Loss; Diabetes Mellitus, Type 2 | interventions — Gastric Bypass

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lifestyle Cohort (Active Comparator): Participants Undergoing Behavioral Weight Loss Program
  Interventions: Behavioral: Behavioral Weight Loss Program
- Surgical Cohort (Active Comparator): Participants Scheduled for Roux-en-Y Gastric Bypass Surgery
  Interventions: Procedure: Roux-en-Y Gastric Bypass or Sleeve Gastrectomy
- Healthy Weight Control Cohort (No Intervention): Healthy Weight Controls With No Intervention

INTERVENTIONS:
Behavioral: Behavioral Weight Loss Program — Behavioral Weight Loss Program is a modified version of the Diabetes Prevention Program (DPP).
  Arms: Lifestyle Cohort
Procedure: Roux-en-Y Gastric Bypass or Sleeve Gastrectomy — Subjects undergoing Roux-en-Y Gastric Bypass or Sleeve Gastrectomy with their own surgical team
  Arms: Surgical Cohort

SUMMARY:
Patients and clinicians need better options to prevent the weight regain that almost universally follows a weight loss intervention. In lay terms, a new, higher "set point" seems to occur after people gain weight. Evidence from some research studies reinforces these observations, showing that processes of energy homeostasis vigorously defend the higher level of adiposity for years, if not permanently. Only bariatric surgery appears to "re-set" to a lower level of adiposity. No clear mechanism has been elucidated to date that explains these phenomena. The current proposal endeavors to address this crucial scientific gap by translating preclinical data into human studies testing novel mechanistic hypotheses. Prior studies in rodents show that a high-fat diet causes inflammation and a cellular response, known as gliosis, within hypothalamic regions regulating energy balance and glucose homeostasis. Evidence further suggests that gliosis might play a pathogenic role in obesity and type 2 diabetes mellitus (T2D) because its development precedes weight gain and impaired glucose homeostasis and its inhibition improves metabolic health. Importantly, gliosis is detectable in mice and humans by magnetic resonance imaging (MRI). Using MRI, the investigators discovered the first evidence of gliosis in obese humans and went on to show associations of gliosis with insulin resistance in humans, independent of the level of adiposity. New findings suggest that people with T2D have more extensive gliosis than is seen in nondiabetic obese subjects. Further findings reveal that gliosis improves, but is not completely reversed, 8 mo. after Roux-en-Y gastric bypass (RYGB) surgery in T2D patients. It remains unknown whether gliosis improves similarly when weight loss occurs by lifestyle change or if the efficacy and durability of weight loss via bariatric surgery is partially explained by its ability to reverse gliosis via an as yet unknown mechanism of action. We therefore propose three studies in humans to discover 1) if hypothalamic gliosis is reversed by a standard behavioral weight loss intervention, 2) if the extent of gliosis predicts successful weight loss during, or weight regain after, behavioral weight loss, and 3) the time course of improvement in gliosis after RYGB and the relation of its improvement to the short- and long-term efficacy of RYGB. Future research would define dietary, environmental, or other risk factors for the development of hypothalamic gliosis in humans. Achieving a better understanding of the role of the brain in obesity and its treatment could open new avenues for research, intervention, and prevention.

ELIGIBILITY:
Inclusion Criteria:

* Aged 25-64 years
* Behavioral Weight Loss (BWL) & Surgical Weight Loss (SWL) (Roux-en-Y Gastric Bypass (RYGB) or Sleeve Gastrectomy): BMI 30- <56 kg/m²
* RYGB and Sleeve Gastrectomy: eligible for RYGB or Sleeve Gastrectomy and not undergoing revision or reoperation
* Healthy Weight Controls (HWC): BMI 18.5-24.9 kg/m²

Exclusion Criteria:

* Poorly controlled hypertension or coronary artery disease, or chronic disease (e.g. cancer, multiple sclerosis, autoimmune disease, rheumatic disease) Blood Pressure > 160/100 mmHG Heart Rate > 110 bpm
* Chronic kidney disease (GFR <60 mL/min/1.73 m2),
* Presence of cirrhosis (Nonalcoholic Fatty Liver Disease (NALFD)/Nonalcoholic Steatohepatitis (NASH) are acceptable),
* Previous or planned (during the study period) obesity treatment with surgery (planned surgery ok for the SWL group) or a weight loss device. However, the following are allowed: (1) liposuction and/or abdominoplasty, if performed > 1 year before screening, (2) lap banding, if the band has been removed > 1 year before screening, (3) intragastric balloon, if the balloon has been removed > 1 year before screening or (4) duodenal-jejunal bypass sleeve, if the sleeve has been removed > 1 year before screening,
* A1c > 8.5% in Bariatric group; A1c ≥ 6.5% for BWL and HWC groups,
* Current use of insulin (insulin ok for Surgical Weight Loss group, also called SWL), DPP-4 inhibitors, thiazolidinediones or medications known to alter metabolic function (e.g. atypical antipsychotics, corticosteroids),
* Pregnancy or breastfeeding,
* MRI contraindications (e.g. implanted metal, claustrophobia), or unable to have MRI or fit in MRI scanner
* Current smoking/daily use of nicotine containing products (cigarettes, e-cigarettes, vaping or other nicotine containing products) or heavy alcohol use,
* Weight >450 pounds (iDXA limit),
* Weight-reduced from lifetime maximum weight by >16%,
* Weight not stable over past 3 months (±10%),
* T2D (for BWL or HWC),
* Inability to participate in a weight loss program (BWL)
* History of eating disorder or current eating disorder, currently enrolled in a weight loss program (ok for the SWL group provided weight stability and lifetime weight-reduced maximum conditions are met) or taking medications to lose weight
* Severe food allergies
* Any condition that the study physician determines to be unsafe for participation

Ages: 25 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 112 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2025-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Schur, MD, MS, Principal Investigator — University of Washington
Locations (1):
- University of Washington - South Lake Union, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lifestyle Cohort | Surgical Cohort | Healthy Weight Control Cohort
Started | 72 | 13 | 27
Completed | 52 | 9 | 21
Not Completed | 20 | 4 | 6
Not completed — Withdrawal by Subject | 7 | 2 | 1
Not completed — Lost to Follow-up | 13 | 1 | 4
Not completed — Physician Decision | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lifestyle Cohort | Surgical Cohort | Healthy Weight Control Cohort | Total
Number analyzed (Participants) | 72 | 13 | 27 | 112
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.3 (10.8) | 39.3 (10.9) | 34.7 (11.0) | 40.2 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 12 | 17 | 82
  Male | 19 | 1 | 10 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 0 | 5 | 11
  Not Hispanic or Latino | 65 | 13 | 22 | 100
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 5 | 1 | 5 | 11
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 3 | 0 | 1 | 4
  White | 56 | 9 | 20 | 85
  More than one race | 7 | 3 | 1 | 11
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 72 | 13 | 27 | 112
Weight [Mean (Standard Deviation); unit: kilograms] | 105.4 (17.4) | 105.0 (11.9) | 65.0 (10.0) | 95.5 (23.1)
BMI [Mean (Standard Deviation); unit: kg/m2] | 37.3 (5.4) | 40.4 (4.2) | 22.2 (1.8) | 34.0 (8.2)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Weight From Baseline
Time Frame: During 6 Month Behavioral Weight Loss Program
Population: This analysis considers participants with available weight data at baseline and 6-months (end of treatment).
Measure: Mean (Standard Error); unit: percentage change from baseline
Arm/Group | Lifestyle Cohort | Surgical Cohort | Healthy Weight Control Cohort
Number analyzed (Participants) | 56 | 11 | 18
percentage change from baseline | -6.1 (0.8) | -21.2 (1.9) | 1.2 (0.7)
Statistical Analysis 1: Comparison: Lifestyle Cohort vs Surgical Cohort vs Healthy Weight Control Cohort; Test type: Superiority; p < 0.001, ANOVA

2. Primary Outcome: Weight Regain
Description: Change in Weight (kg) during 12 month follow-up period
Time Frame: During 12-Month Follow-Up After Intervention
Population: This analysis considers participants with available data at the end of treatment visit (6-month visit) and 12-months later (18-month visit).
Measure: Mean (Standard Error); unit: change in kg during 12M follow up
Arm/Group | Lifestyle Cohort | Surgical Cohort | Healthy Weight Control Cohort
Number analyzed (Participants) | 45 | 9 | 16
change in kg during 12M follow up | 0.7 (2.1) | -1.8 (2.2) | 0.1 (0.7)
Statistical Analysis 1: Comparison: Lifestyle Cohort vs Surgical Cohort vs Healthy Weight Control Cohort; Test type: Superiority; p = 0.85, ANOVA

ADVERSE EVENTS:
Time Frame: About 18 months.
Arm/Group | Lifestyle Cohort | Surgical Cohort | Healthy Weight Control Cohort
All-Cause Mortality (participants affected / at risk) | 0/72 | 0/13 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/72 | 0/13 | 0/27
Other Adverse Events (participants affected / at risk) | 0/72 | 0/13 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2023-04-19): https://cdn.clinicaltrials.gov/large-docs/87/NCT03578887/Prot_000.pdf
  • Statistical Analysis Plan (2025-06-09): https://cdn.clinicaltrials.gov/large-docs/87/NCT03578887/SAP_001.pdf
  • Informed Consent Form (2022-08-22): https://cdn.clinicaltrials.gov/large-docs/87/NCT03578887/ICF_002.pdf